CLINICAL TRIAL: NCT05997511
Title: Leveraging Community Health Workers to Combat Health Misinformation in Haiti, Malawi, and Rwanda
Brief Title: Leveraging Community Health Workers to Combat COVID-19 and Mental Health Misinformation in Haiti, Malawi, and Rwanda
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard Medical School (HMS and HSDM) (Other)
Collaborators: Partners in Health (Other)
Responsible Party: Principal Investigator, Bethany Hedt-Gauthier, Principal Investigator, Harvard Medical School (HMS and HSDM)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB22-1339
Record Dates: First submitted 2023-07-22; First posted 2023-08-18 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Mental Health; COVID-19; Misinformation
Keywords: COVID-19; Mental Health; Misconception; Community Health Workers (CHWs)
MeSH Terms: conditions — Psychological Well-Being; COVID-19; Communication

STUDY DESIGN:
Intervention Model Description: Our study will use a cluster- randomized design with two active arms - one arm targeting COVID-19-related misinformation and a second arm targeting misinformation related to mental health.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COVID-19 (Other): Behavioral (SMS) Intervention
  Interventions: Behavioral: Card-Sorting Activity (Pre-intervention design); Behavioral: SMS Crafting (Pre-intervention design); Behavioral: SMS Messaging
- Mental Health (Other): Behavorial (SMS) Intervention
  Interventions: Behavioral: Card-Sorting Activity (Pre-intervention design); Behavioral: SMS Crafting (Pre-intervention design); Behavioral: SMS Messaging

INTERVENTIONS:
Behavioral: Card-Sorting Activity (Pre-intervention design) — Study team members within each country will free list misinformation or misconceptions that they commonly encounter in clinical practice or daily life. Each item will be used to create paired cards - one containing the misinformation and a second containing the corresponding correct information. During qualitative interviews, we will ask CHWs to participate in a series of card sorting activities, which is a participatory research method that can inform the design of health interventions.
Behavioral: SMS Crafting (Pre-intervention design) — A two-person team consisting of one local communication expert and one clinician will draft clinically correct, easy-to-understand SMS messages designed to counter identified misinformation. We will draft messages that use various styles and use cognitive interviewing with CHWs to assess their understanding of and responses to each style. The final messages used in our intervention will be determined by CHW preference.
Behavioral: SMS Messaging — Final messages will be sent via SMS to all CHWs working in our study area. CHWs will also be provided with contact information for a helpline staffed by a local team member who can answer follow-up questions in the local language.
  Other Names: text messaging

SUMMARY:
Partners In Health (PIH), in collaboration with Harvard Medical School, aims to develop and evaluate an SMS-based intervention for Community Health Workers (CHWs) to combat COVID-19 and mental health-related misinformation in Haiti, Rwanda, and Malawi. The study involves three aims: identifying locally relevant misinformation through a card-sorting exercise with CHWs, developing targeted messages through cognitive interviewing, and evaluating the effectiveness of SMS-based educational message dissemination via a randomized controlled trial. The evaluation will assess the impact on public health practices, knowledge and attitudes among CHWs, and knowledge and attitudes among community members.

DETAILED DESCRIPTION:
The intervention will involve sending SMS messages to randomized CHWs, addressing either COVID-19 or mental health misinformation. CHWs will have access to a helpline for further support and can provide feedback to refine the messaging. The evaluation will use a time series analysis to measure changes in COVID-19 vaccine administration, mental health service utilization, CHWs' knowledge and attitudes, and community members' knowledge and attitudes. The study aims to empower CHWs with accurate information, improve public health practices, and ultimately contribute to better health outcomes in the communities served by PIH. Rwanda and Haiti CHWs will receive the messages for 12 months, but Malawi CHWs will receive the messages for 6 months due to a CHW transition in country.

ELIGIBILITY:
The intervention will be assigned at the unit of the CHWs. These individuals will also be eligible for the CHW longitudinal cohort.

Inclusion Criteria:

* CHWs affiliated with PIH Rwanda, Malawi, or Haiti
* 18+ years of age.

Exclusion Criteria:

- Less than 18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5109 (Actual)
Dates: Start 2023-11-27 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Number of Mental Health Visits/ Consultations Completed Monthly at Health Facilities | 24 months
  Mental health service utilization will be measured using routinely collected data measured monthly at the health facility level
Number of Patients who Sought Care from Mental Health Services Monthly at Health Facilities | 24 months
  Mental health service utilization will be measured using routinely collected data measured monthly at the health facility level
Number of COVID-19 Vaccine Doses Administered Monthly at Health Facilities (if available) | 24 months
  COVID-19 Vaccine administration will be measured using routinely collected data measured monthly at the health facility level

SECONDARY OUTCOMES:
Qualitative Interviews | Before, after 6 months of the intervention, and after 12 months of the intervention (only in Rwanda & Haiti)
  In-depth qualitative interviews will occur before, during, and after the dissemination of messages. Prior to the message dissemination we will contact between 10-15 randomly selected CHWs per country and provide them with draft messages. Although the content of all messages will be determined by the results of the card sorting exercise, the style of the messages will vary. We will use cognitive interviewing techniques to understand how CHWs interpret each message and ask them to provide their preferences on messaging style. During subsequent qualitative sessions at midline and endline, we will ask up to ten CHWs to provide feedback on the messages that they actually received during the intervention.
Longitudinal Cohort Surveys | Before, after 6 months of the intervention, and after 12 months of the intervention (only in Rwanda & Haiti)
  In each country, we will also select a random sample of 175 CHWs to participate in in a longitudinal cohort consisting of a quantitative questionnaire administered before, during, and after the intervention. During our survey, we will assess both COVID-19 related outcomes (CHWs' knowledge about COVID-19, vaccination status, and intention to vaccinate) and mental health-related outcomes (CHWs' knowledge about and stigmatization of mental illness). After the start of the intervention, we will also ask CHWs to self-report whether they have received our messages or used our helpline, and we will seek to verify this information by direct observation of text messages or outgoing calls on their phone.
Cross-Sectional Survey | Before the intervention and after 12 months of the intervention (only in Rwanda & Haiti)
  a repeated cross-sectional survey of community members

CONTACTS AND LOCATIONS:
Locations (3):
- Zanmi Lasante, Cangé, Haiti
- Partners in Health- Malawi, Neno, Malawi
- Partners in Health- Rwanda, Kigali, Rwanda

IPD SHARING:
Plan to Share IPD: No